CLINICAL TRIAL: NCT05829395
Title: The Effect of Metaverse-based Education on Nursing Students' Learning Motivation and Academic Achivement
Brief Title: The Use of Metaverse in Nursing Education
Acronym: metaverse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Ayşe Aydınlı, Research Asistant, RN, MsN, PhD, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SuleymanSDU
Record Dates: First submitted 2023-04-10; First posted 2023-04-25 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Nursing Student
Keywords: Nursing student; Motivation; metaverse; Academic achievement

STUDY DESIGN:
Intervention Model Description: This study will be conducted as a randomized controlled experimental study in order to determine the effect of nursing process teaching in the metaverse environment on the learning motivation and academic achievement of nursing students. this study will be conducted from March 2023 to April 2023 in the nursing department of a university. The sample consisted of 42 students who volunteered to participate in the research and met the inclusion criteria. Scales and Forms to be used in the Study; Personal Information Form, The Instructional Materials Motivation Scale, and Academic Success Assessment (Quiz)
Who Masked: Participant
Masking Description: With the simple randomization method, students will be assigned to the experimental and control groups. But students will not know which group is the experimental group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention Group (Experimental): Starting from the week following the pre-test application, online training will continue according to the Metaverse-based for a total of 3 weeks, two hours a week, for the intervention group. At the end of the 3 weeks, the Instructional Materials Motivation Scale and Academic Success Assessment (Quiz) will be re-administered as a post-test.
  Interventions: Other: metaverse- based education
- Control Group (No Intervention): The subjects were explained by the instructor with the traditional e-teaching method. The subjects will be explained by the instructor with the traditional e-teaching method and as in the intervention group, the lectures were conducted online for two hours a week for 3 weeks. At the end of the 3 week, the post-tests of the Instruvtional Materials Motivation Scale and Academic Success Assessment (Quiz) will be apply in the control group simultaneously with the intervention group.

INTERVENTIONS:
Other: metaverse- based education — The nursing process course will be conducted in a metaverse environment. A virtual classroom is designed in the metaverse space for the execution of this course.
  Starting from the week following the pre-test application, online training will continue according to the Metaverse-based for a total of 3 weeks, two hours a week, for the intervention group. At the end of the 3 weeks, the Instructional Materials Motivation Scale and Academic Success Assessment (Quiz) will be re-administered as a post-test.
  Arms: İntervention Group

SUMMARY:
This study will be conducted as a randomized controlled experimental study in order to determine the effect of nursing process teaching in the metaverse environment on the instructional materials motivation and academic achievement of nursing students. this study will be conducted from March 2023 to April 2023 in the nursing department of a university. The sample consisted of 42 students who volunteered to participate in the research and met the inclusion criteria.

DETAILED DESCRIPTION:
This study will be conducted as a randomized controlled experimental study to determine the effect of nursing process teaching in the metaverse environment on the instructional materials motivation and academic achievement of nursing students. The nursing process course will be conducted in a metaverse environment. A virtual classroom is designed in the metaverse space for the execution of this course. This study will be conducted from March 2023 to April 2023 in the nursing department of a university. The sample consisted of 42 students who volunteered to participate in the research and met the inclusion criteria. Scales and Forms to be used in the Study; Personal Information Form, The Instructional Materials Motivation Scale, and Academic Success Assessment (Quiz). With the simple randomization method, students will be assigned to the experimental and control groups. But students will not know which group is the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* Having volunteered to participate in the study
* Being a first-year nursing student
* Taking the course nursing process
* Students with unlimited access to the internet and computer

Exclusion Criteria:

* Not having volunteered to participate in the study
* Students who do not taking and continuing in the nursing process course

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Personal Information Form | one week
  This form was prepared by the researchers to determine some sociodemographic characteristics of the participating students. The form consists of 6 questions regarding characteristics of the students' such as age, gender, and graduated high school.
The Instructional Materials Motivation Scale | 3 weeks
  Investigators uses the five-point Likert scale: "strongly agree," "agree," "neutral," "disagree," and "strongly disagree". The original IMMS consisted of 36 questions and four dimensions (attention, relevance, confidence, and satisfaction). The Cronbach's α of the overall questionnaire is 0.96 and the Cronbach's α for each of the sub-dimensions ranges between 0.81 and 0.92. A Turkish version of IMMS was constructed from 24-items.
Academic Success Assessment (Quiz) | 3 weeks
  It is a 16 multiple-choice exam created by the researcher to measure the success of the students in the Nursing Process course. This exam lasted 18 minutes. Each question is worth 6.25 points.

CONTACTS AND LOCATIONS:
Overall Officials: Esin Çetinkaya Uslusoy, Study Chair — Suleyman Demirel University
Locations (1):
- Suleyman Demirel University, Isparta, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao J, Lu Y, Zhou F, Mao R, Fei F. Systematic Bibliometric Analysis of Research Hotspots and Trends on the Application of Virtual Reality in Nursing. Front Public Health. 2022 May 19;10:906715. doi: 10.3389/fpubh.2022.906715. eCollection 2022. PMID 35664095
- [Background] Ahuja AS, Polascik BW, Doddapaneni D, Byrnes ES, Sridhar J. The Digital Metaverse: Applications in Artificial Intelligence, Medical Education, and Integrative Health. Integr Med Res. 2023 Mar;12(1):100917. doi: 10.1016/j.imr.2022.100917. Epub 2022 Dec 22. No abstract available. PMID 36691642
- [Background] Bhugaonkar K, Bhugaonkar R, Masne N. The Trend of Metaverse and Augmented & Virtual Reality Extending to the Healthcare System. Cureus. 2022 Sep 12;14(9):e29071. doi: 10.7759/cureus.29071. eCollection 2022 Sep. PMID 36258985
- [Result] Ali S, Abdullah, Armand TPT, Athar A, Hussain A, Ali M, Yaseen M, Joo MI, Kim HC. Metaverse in Healthcare Integrated with Explainable AI and Blockchain: Enabling Immersiveness, Ensuring Trust, and Providing Patient Data Security. Sensors (Basel). 2023 Jan 4;23(2):565. doi: 10.3390/s23020565. PMID 36679361